CLINICAL TRIAL: NCT05422287
Title: The Effect of Using a Thermomechanical Stimulation Device and Virtual Reality Glasses During Peripheral Intravenous Catheter Administration on Pain and Patient Satisfaction in Adult Patients
Brief Title: Effect of Thermomechanical Stimulation Device and Virtual Reality Glasses During Peripheral Intravenous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ebru Erek Kazan, Assist.Prof.Dr., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/76
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Catheterization
Keywords: Nursing; pain; patient satisfaction; peripheral intravenous catheterization; thermomechanical stimulation; virtual reality
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (VRG) Group (Experimental): The participants in this group were started to watch videos by wearing virtual reality glasses about 2 minutes before the catheterization process was started and the process was continued until the end. Then, catheterization was performed by detecting the tourniquet by the emergency department nurse. Upon completion of the catheterization procedure, VRG was removed from the procedure area by the researcher. This process took an average of 5 minutes. After the procedure was completed, the pain and satisfaction status of the patients were scored on the VAS by the same nurse.
  Interventions: Other: Virtual Reality Glasses
- Thermomechanical Stimulation Device (Buzzy ®) Group (Experimental): 1 minute before starting the catheterization procedure in this group, a cold and vibration application was placed in the operation area by the researcher using the apparatus of the Buzzy ® device and started. The procedure was performed after evaluating the vein and determining the appropriate right or left arm. At the end of this time, the Buzzy ® has been shifted approximately 5 cm above the processing zone. Then, catheterization was performed. Upon completion of the catheterization procedure, Buzzy ® was removed from the procedure area by the researcher. This process took an average of 4 minutes. After the procedure was completed, the pain and satisfaction status of the patients were scored on the VAS by the same nurse.
  Interventions: Other: Thermomechanical Stimulation Device
- Control group (No Intervention): Peripheral intravenous catheterization was performed by the same emergency department nurse in accordance with the procedure. The process took an average of 3 minutes. There was no application to the patients in the control group except for the standard procedure. After the procedure was completed, the pain and satisfaction status of the patients were scored on the VAS by the same nurse.

INTERVENTIONS:
Other: Virtual Reality Glasses — Group 1
  Other Names: VRG
  Arms: Virtual Reality Glasses (VRG) Group
Other: Thermomechanical Stimulation Device — Group 2
  Other Names: Buzzy
  Arms: Thermomechanical Stimulation Device (Buzzy ®) Group

SUMMARY:
The study was conducted as a randomized controlled experimental study to determine the effect of Thermomechanical Stimulation Device (Buzzy®) and Virtual Reality Goggles (VRG) applied during peripheral intravenous catheterization (PIC) on pain and patient satisfaction in adult patients.

DETAILED DESCRIPTION:
The research was carried out at the Emergency Department of the Etimesgut Şehit Sait Ertürk State Hospital in Ankara from April 2021 to February 2022. The sample of the study consisted of 126 adult patients. The patients were divided into three groups by randomization method. VRG was applied to the first group, Buzzy to the second group and the control group which was the third group using the standard procedure. Before the procedure of PIC, "Introductory Characteristics Form for Patients" was prepared by the researcher containing the sociodemographic characteristics of the participants (gender, marital status, age, educational status, etc. as such). This form was filled out by asking the patient by face-to-face interview method. After catheterization, the "Visual Comparison Scale for Pain" was used by the nurse practitioner to determine the pain of the patients and the "Visual Comparison Scale for Satisfaction" was used to determine the satisfaction status of the patients regarding the application to be performed. It is expected that pain and patient satisfaction scores in groups where a VRG and Buzzy® were used during PIC in adult patients will result more positively than in the control group. It is thought that the results obtained from the research will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Shold be a volunteer to participate in the research
* Should be in the age of between 18-65 years old
* Should not use drugs that will have an analgesic effect in the last 24 hours before admission
* Should have successful of the first intravenous catheterization attempt
* Absence of any psychiatric illness
* Absence of any oncology and hematology disease
* Should have the ability to read and write in Turkish,
* Absence of vision, hearing and perception problems
* Should not have a febrile illness at the time of applications
* Should not have thin and damaged vascular structure
* Absence of a history of fainting during blood removal
* Should be conscious, fully oriented and cooperative, and open to communication

Exclusion Criteria:

* Failure of the first attempt to administer intravenous catheterization
* The unwillingness of the patient to continue the research
* Removing the virtual reality glasses before and during the procedure
* Discontinuing of Buzzy ® before and during the procedure
* Deterioration of the patient's health status during the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Pain of the patient during the peripheral intravenous catheterization | 6 month
  In the study, Visual Analog Scale (VAS) was used to evaluate the pain of the patients. There is a 10 cm ruler on this scale. Patients were asked to rate the pain felt during the procedure on a 10 cm ruler. This scoring was done with a number between 1 and 10. The patient gave a score of "0" if he does not feel pain and "10" if he feels unbearable pain. After the completion of the procedure, the patients were asked to rate the pain they felt during catheterization on a visual comparison scale. At the end of the research, the scale results will be compared and evaluated for all three groups.
Satisfaction of the patients about intervention during the peripheral intravenous catheterization | 6 month
  In the study, another visual comparison scale was used to determine the satisfaction levels of the patients regarding the application to be made. After the completion of the procedure, the patients were asked to rate their satisfaction with the procedure on the Visual Analog Scale (VAS). The scale was scored between 1 and 10, "0" was evaluated as ''I am not satisfied at all'', "10" was evaluated as ''I am very satisfied''. At the end of the research, the scale results will be compared and evaluated in three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Züleyha Setenay Serin, MsN, Principal Investigator — Ankara Yildirim Beyazit University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Yildirim Beyazit University, Faculty of Health Sciences, Department of Nursing, Ankara, Cubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serin ZS, Kazan EE. The Effect of Using Thermomechanical Stimulation and Virtual Reality Glasses During Peripheral Intravenous Catheterization on Pain and Patient Satisfaction: A Randomized Controlled Trial. J Emerg Nurs. 2025 Sep;51(5):925-935. doi: 10.1016/j.jen.2025.04.005. Epub 2025 May 26. PMID 40418199